CLINICAL TRIAL: NCT03030547
Title: Erişkin Kas hastalıklarında Fiziksel Aktivite Ile ilişkili faktörlerin Belirlenmesi
Brief Title: Identification of Factors Associated With Physical Activity Levels in Adult Muscle Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Fatma Ayvat, Principal Investigator, Research Assistant, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GO 14/617
Record Dates: First submitted 2017-01-15; First posted 2017-01-25 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Muscle Disease
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Muscle Disease Group (Experimental): Adult patients with muscle diseases diagnosed by neurologist, will wear SenseWear activity monitor for 5 days
  Interventions: Device: SenseWear activity monitor
- Healthy Individuals Group (Active Comparator): Healthy individuals with similar demographic characteristics as adult patients with muscle diseases, will wear SenseWear activity monitor for 5 days
  Interventions: Device: SenseWear activity monitor

INTERVENTIONS:
Device: SenseWear activity monitor — Individuals will wear SenseWear activity monitors on right triceps muscle for 5 days. The data stored on the device will be recorded in computer using the software. Individuals will be given information of the resulting data (total number of steps, total energy expenditure, the number of daily steps and energy expenditure, physical activity duration in different intensity).

SUMMARY:
To evaluate physical activity levels and factors associated with physical activity levels in adult patients with muscle diseases.

DETAILED DESCRIPTION:
The same protocol will be applied all of the patients and healthy subjects. Individuals will be informed in detail about the study and demographic and physical properties will recorded after receiving approval. Evaluation programme that consisting of pain, fatigue, falls, activity limitations, quality of life, muscle strength assessment and functional assessment will be applied. After the evaluation, individuals will be given detailed information on the use of SenseWear activity monitors. Individuals will wear SenseWear activity monitors on right triceps muscle for 5 days. The data stored on the device will be recorded in computer using the software. Individuals will be given information of the resulting data (total number of steps, total energy expenditure, the number of daily steps and energy expenditure, physical activity duration in different intensity). Physical activity levels will be assessed by subjective aspects of physical activity questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of muscle diseases
* Adult patients with muscle diseases who are able to walk independently

Exclusion Criteria:

* Clinical diagnosis of systemic problems
* Any orthopedic problems that will affect the performance of the physical activity
* Clinical diagnosis of neurological disease other than muscle disease
* Clinical diagnosis of cognitive impairment
* Individuals who underwent surgery in the last 6 month

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Energy expenditure on SenseWear Activity Monitor | 5 days
  The SenseWear software calculates energy expenditure based on a proprietary algorithm that incorporates subject height, weight, age, and sex which are entered prior to data analysis as well as the various measurements (two-axis accelerometry, galvanic skin response, heat flux, skin and near-body temperature).
Number of steps on SenseWear Activity Monitor | 5 days
  The SenseWear software calculates number of steps based on a proprietary algorithm that incorporates subject height, weight, age, and sex which are entered prior to data analysis.

SECONDARY OUTCOMES:
International Physical Activity Scale (IPAQ) | 10 minutes
  27 item self-reported measure of physical activity for use with individual adult patients aged 15 to 69 years old. The IPAQ can be used clinically and in population research that compares physical activity levels between populations internationally. Duration (minutes) and frequency (days) of physical activity in the last 7 days is measured in domains of: Job-related, transportation, housework, house maintenance, caring for family, recreation, sport, leisure-time and time spent sitting. Overall score calculated using responses to all questions (Score is obtained by multiplying duration and frequency for each question) and total MET-min/week score obtained.
Visual Analog Scale | 2 minutes
  10 cm line anchored at both ends with words descriptive of the maximal and minimal extremes of the pain being measured. Individuals mark their pain intensity on a line numbered 0-10.
Fatigue Severity Scale | 5 minutes
  The 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders.. The items are scored on a 7 point scale with 1 = strongly disagree and 7= strongly agree. The minimum score = 9 and maximum score possible = 63. Higher the score = greater fatigue severity.
ACTIVLIM questionaire | 5 minutes
  The ACTIVLIM questionnaire explores difficulties of performing daily activities that required the use of upper limbs or/and the use of lower limbs. The adult patients and the parents of affected children fill in either the adult form or the child form of the questionnaire. They are asked to provide their perceived difficulty in performing each activity using a three-level scale: impossible (0), difficult (1), easy (2). Each activity must be completed without technical or human assistance.
Medical Outcomes Short-Form Health Survey | 10 minutes
  The SF-36 is a generic patient-reported outcome measure aimed at quantifying health status, and is often used as a measure of health-related quality of life. The SF-36 is a 36-item questionnaire that measures the physical and mental health constructs of health status. These constructs are measured through 8 subscales. The physical component (PCS) is made up of physical functioning (PF), role-physical (RP), bodily pain (BP), and general health (GH). The Mental component (MCS) is made up of vitality (VT), social functioning (SF), role-emotional (RE), and mental health (ME). Each of the 36 items is answered using a Likert-type scale and a 4-week recall period, with a total score of 0-100 possible. A higher score indicates better health status.
Hand Held Dynamometry | 20 minutes
  A quantitative and objective method for assessment of muscular strength using a portable hand held dynamometer. "Break Test" option is used in the study. "Break Test" where the tester applies a force to just overcome the strength of the person being tested, producing an eccentric muscular contraction and scored using force production in Newtons. 3 maximum voluntary isometric contractions are completed and scores summed.
Six Minutes Walk Test | 10 minutes
  Assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance. Walk of cover as far a distance as possible over 6 minute. Assistive devices can be used but kept consistent from test to test. Individual should be able to ambulate without physical assistance.
Timed Up and Go Test | 2 minutes
  Assesses mobility, balance, walking ability, and fall risk. The patient sits in the chair with his/her back against the chair back. On the command "go", the patient rises from the chair, walks 3 meters at a comfortable and safe pace, turns, walks back to the chair and sits down. Timing begins at the instruction "go" and stops when the patient is seated. Patient must use the same assistive device each time he/she is tested to be able to compare scores. 3 trials are completed and scores summed.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Ayvat, Msc, Principal Investigator — Hacettepe University; Muhammed Kılınç, Assoc Prof, Principal Investigator — Hacettepe University; Sibel Aksu Yıldırım, Prof, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McDonald CM. Physical activity, health impairments, and disability in neuromuscular disease. Am J Phys Med Rehabil. 2002 Nov;81(11 Suppl):S108-20. doi: 10.1097/00002060-200211001-00012. PMID 12409816
- [Result] McCrory MA, Kim HR, Wright NC, Lovelady CA, Aitkens S, Kilmer DD. Energy expenditure, physical activity, and body composition of ambulatory adults with hereditary neuromuscular disease. Am J Clin Nutr. 1998 Jun;67(6):1162-9. doi: 10.1093/ajcn/67.6.1162. PMID 9625089
- [Result] Kilmer DD, Wright NC, Aitkens S. Impact of a home-based activity and dietary intervention in people with slowly progressive neuromuscular diseases. Arch Phys Med Rehabil. 2005 Nov;86(11):2150-6. doi: 10.1016/j.apmr.2005.07.288. PMID 16271563
- [Result] Mulligan HF, Hale LA, Whitehead L, Baxter GD. Barriers to physical activity for people with long-term neurological conditions: a review study. Adapt Phys Activ Q. 2012 Jul;29(3):243-65. doi: 10.1123/apaq.29.3.243. PMID 22811565
- [Result] Scheers T, Philippaerts R, Lefevre J. Variability in physical activity patterns as measured by the SenseWear Armband: how many days are needed? Eur J Appl Physiol. 2012 May;112(5):1653-62. doi: 10.1007/s00421-011-2131-9. Epub 2011 Aug 28. PMID 21874552
- [Result] Saglam M, Arikan H, Savci S, Inal-Ince D, Bosnak-Guclu M, Karabulut E, Tokgozoglu L. International physical activity questionnaire: reliability and validity of the Turkish version. Percept Mot Skills. 2010 Aug;111(1):278-84. doi: 10.2466/06.08.PMS.111.4.278-284. PMID 21058606
- [Result] Brinkmann JR. Comparison of a hand-held and fixed dynamometer in measuring strength of patients with neuromuscular disease. J Orthop Sports Phys Ther. 1994 Feb;19(2):100-4. doi: 10.2519/jospt.1994.19.2.100. PMID 8148862
- [Result] Armutlu K, Korkmaz NC, Keser I, Sumbuloglu V, Akbiyik DI, Guney Z, Karabudak R. The validity and reliability of the Fatigue Severity Scale in Turkish multiple sclerosis patients. Int J Rehabil Res. 2007 Mar;30(1):81-5. doi: 10.1097/MRR.0b013e3280146ec4. PMID 17293726
- [Result] Price DD, Bush FM, Long S, Harkins SW. A comparison of pain measurement characteristics of mechanical visual analogue and simple numerical rating scales. Pain. 1994 Feb;56(2):217-226. doi: 10.1016/0304-3959(94)90097-3. PMID 8008411
- [Result] Vandervelde L, Van den Bergh PY, Goemans N, Thonnard JL. ACTIVLIM: a Rasch-built measure of activity limitations in children and adults with neuromuscular disorders. Neuromuscul Disord. 2007 Jun;17(6):459-69. doi: 10.1016/j.nmd.2007.02.013. Epub 2007 Apr 11. PMID 17433675
- [Result] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Result] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Result] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914